CLINICAL TRIAL: NCT05162612
Title: Anatomo-radiological Study on Semilunar Line as Risk Factor fo Diastasis Recti Abdominis
Acronym: Semilunare
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marta Cavalli (Other)
Responsible Party: Sponsor-Investigator, Marta Cavalli, co-Investigator, researcher in General Surgery, University of Insubria, Surgeon in Istituto Clinico Sant'Ambrogio - Centro di Ricerca di Alta Specializzazione sulla Patologia della Parete Addominale e sulla Chirurgia Riparativa delle Ernie Addominali, Università degli Studi dell'Insubria
Organization: Università degli Studi dell'Insubria (Other)
Other Study IDs: Semilunare
Record Dates: First submitted 2021-11-16; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Diastasis Recti and Weakness of the Linea Alba
Keywords: diastasis recti abdominal; abdominal wall hernia; semilunar line; internal oblique muscle; external oblique muscle; transversal muscle
MeSH Terms: conditions — Diastasis Recti And Weakness Of The Linea Alba; Hernia, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: abtominal CT — standard basic Abdominal Ct scan

SUMMARY:
Multicenter cross-sectional observational study with the aim of investigating the prevalence of diastasis recti abdominis in adults and identifying its risk factors.

Secondary outcoms:

* identify the presence of possible risk factors for diastasis recti abdominis
* evaluate the insertion of the aponeurosis of the internal oblique muscle in the semilunar line in abdominal CT in a large series of patients
* investigate the prevalence of the presence of only the posterior insertion of the internal oblique aponeurosis
* evaluate the correlation of the presence of only the posterior lamella with the diastasis recti abdominia and with the pathology of the abdominal wall (ventral and/or incisional hernia)
* evaluate the correlation between diastasis and other anatomo-radiological findings, such as the thickness of the rectus muscles and the distance between the lateral edge of the rectus muscles with the medial edges of the lateral abdominal muscles (external oblique, internal oblique and transverse)
* evaluate the variability of the results

DETAILED DESCRIPTION:
As usually described, at the lateral margin of the rectus sheath, the lateral muscles aponeurosis joins themselves in the semilunar line. The external oblique (EO) aponeurosis constantly passes in front of the rectus muscle (RM), composing the anterior lamina of the sheath. The internal oblique (IO) aponeurosis splits its fibers in an anterior and a posterior layer. The anterior layer joins the fibers of the EO in front of RM to constitute the anterior lamina. But some centimeters below the umbilicus, there is no split in the fibers, and all the aponeurosis of the IO join the EO and transverse aponeurosis in constituting the anterior sheath. The transverse muscle aponeurosis also behaves differently from cranial to caudal. Cranially the fibers constantly remain posterior to the RM and constitutes the deep layer of the sheath, but at a variable level some centimeters below the umbilicus, they go anteriorly will all other flat muscle aponeurosis.

During cadaveric dissections and in a careful evaluation of various CT abdominal wall images, we noted that the IO aponeurosis can join the rectus sheath in two ways: a) splitting its fibers in an anterior and posterior layer, as classically described, or b) joining only the posterior rectus sheath without an anterior layer.

To confirm our hypothesis, we design this multicenter cross-sectional observational study.

Data collection:

For each patient, together principal endpoints, following additional variables will be collected:

* Age
* Sex
* BMI
* Previous abdominal surgical procedures (type and date)
* Diabetes affection
* Number of pregnancies and multiple birth, date of delivery and type of delivery (vaginal or caesarean section)

CT evaluation

A researcher, trained by an expert radiologist, will evaluate the axial image of abdominal standard CT to identify and record:

* the internal oblique aponeurosis insertion in both side: classical double (anterior and posterior) insertion or only posterior insertion
* The inter-recti distance at three regions, including supraumbilical (4,5 cm above the umbilicus), periumbilical and subumbilical (4.5 cm below the umbilicus)
* The thickness and width of both rectus muscles
* The distance between lateral edge of the rectus muscle and the medial edge of the internal oblique muscle
* The distance between lateral edge of the rectus muscle and the medial edge of the external oblique muscle
* The distance between lateral edge of the rectus muscle and the medial edge of the transverse muscle
* Presence of abdominal wall hernia, if any

Definition and classification of DRA According Rath et al. (13) proposal, for subjects younger than 45 years, DRA will be defined as a separation of the two recti more than 1.0 cm above the umbilicus, 2.7 cm at the periumbilicus and 0.9 cm below the umbilicus; for subjects over 45 years, the corresponding values will be 1.5 cm, 2.7 cm and 1.4 cm, respectively. The presence of an inter-recti distance superior to the cut off value in two or three regions (supraumbilical, umbilical and subumbilical) in the same patient will be described as DRA.

Width of the DRA will be defined according Ranney (15) classification: an IRD < 3 cm will be labeled mild diastasis, 3-5 cm IRD moderate diastasis and more than 5 cm severe diastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can undergo CT examination
* Adult patients (men and women, minimum age 18) requiring an abdominal CT scan, for any diagnostic indication
* Signed informed consent for partecipation to the study and for processing of sensitive data
* Filled anamnestic questionnaire

Exclusion Criteria:

* Patients with severe neurological / psychiatric conditions
* Minor patients (age <18 years)
* women with a recent pregnancy or birth (in the last year)
* patients with recent abdominal surgery (within the last six months).

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients requiring a Ct abdominal scan, for any diagnostic indication
Sampling Method: Probability Sample
Enrollment: 987 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2023-09-13 (Estimated)

PRIMARY OUTCOMES:
Prevalence of diastasis | 2 years
  Number of patients presenting diastasis. According Rath et al. proposal, for subjects younger than 45 years, diastasis will be defined as a separation of the two recti more than 1.0 cm at 45mm above the umbilicus, 2.7 cm at the periumbilicus and 0.9 cm at 45 mm below the umbilicus; for subjects over 45 years, the corresponding values will be 1.5 cm, 2.7 cm and 1.4 cm, respectively.

SECONDARY OUTCOMES:
insertion of the internal oblique apneurosis | 2 years
  Accordin our hypothesis the internal oblique aponeurosis can join the rectus sheath in two way: a) splitting its fibers in an anterior and posterior layer, as classically described, or b) joining only the posterior rectus sheath without an anterior layer.
  We will evaluted how many patient presentig a double insertion (anterior and posterior) and how many a single posterior insertion
correlation between diastasis and type of internal oblique insertion | 2 years
  number of patient with single posterior insertion presenting diastasis and number of patient with classic double insertion presentig diastasis
correlation between abdominal wall hernia and type of internal oblique insertion | 2 years
  number of patient with single posterior insertion presenting hernia and number of patient with classic double insertion presentig hernia
correlation between diastasi and other anatomo-radiolpgical findings | 2 years
  the following measures will be taken:
  * tickness of both rectus muscle (mm)
  * width of both rectus muscle (mm)
  * distance (mm) between the laterl edge of retus muscle and the medial edge of external oblique muscle, internal oblique muscle and trasnversus muscle

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Clinico Sant'Ambrogio - Centro di Ricerca di Alta Specializzazione sulla Patologia della Parete Addominale e sulla Chirurgia Riparativa delle Ernie Addominali, Milan
  - Ospedale di Circolo e Fondazione Macchi di Varese, Varese

REFERENCES:
- [Result] Cavalli M, Aiolfi A, Bruni PG, Manfredini L, Lombardo F, Bonfanti MT, Bona D, Campanelli G. Prevalence and risk factors for diastasis recti abdominis: a review and proposal of a new anatomical variation. Hernia. 2021 Aug;25(4):883-890. doi: 10.1007/s10029-021-02468-8. Epub 2021 Aug 6. PMID 34363190